CLINICAL TRIAL: NCT02973880
Title: A Prospective, Multi-center, Controlled, Double-blind Study to Evaluate the Efficacy and Tolerability of a Steroid/Antibiotic Associated Treatment Following Cataract Extraction by Means of Phaco-emulsification
Brief Title: Clinical Study to Evaluate the Efficacy and Tolerability of an Anti-inflammatory/Antibiotic Treatment Following Ocular Cataract Extraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SIFI SpA (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 044-SI; 2016-002138-63 (EudraCT Number)
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Cataract Extraction; Cataract
Keywords: Steroid/antibiotic associated treatment; Phaco-emulsification; Cataract extraction
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Two treatment arms, test group versus active-comparator (control) group, treated in parallel.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All daily study products will be manufactured in indistinguishable single dose plastic vials, labeled in accordance with hour of administration. In accordance with the double-blind design of the study, daily treatment for patients randomized to group A (NETILDEX™ ophthalmic gel), will be of 2 doses of active treatment and 2 doses of indistinguishable placebo. For blinding purposes, Group B (NETILDEX™ eye drops solution) medications labels will consist in an aluminum envelope for each dose of the daily treatment, containing indistinguishable plastic vials of NETILDEX™ eye drops solution. Tertiary packaging (patient's treatment supply) will be a carton box appropriately labeled, containing 16 secondary packages (aluminum envelopes - each envelope containing 5 vials for each treatment time dose), containing enough plastic vials to allow the patient to complete the whole study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NETILDEX™ ophthalmic gel (Experimental): 1 drop of NETILDEX™ (Netilmicin Sulfate 3mg/ml / Dexamethasone Disodium Phosphate 1mg/ml) ophthalmic gel immediately after the surgery then 1 drop twice daily (b.i.d.) from Day 1 until Day 14 after surgery + 1 drop of XANTERGEL™ ophthalmic gel twice daily (b.i.d.) from Day 1 until Day 14 after surgery.
  Bromfenac 0.9 mg/ml 1 drop twice daily (b.i.d.) for 3 days before cataract surgery.
  Interventions: Drug: NETILDEX™ ophthalmic gel
- NETILDEX™ eye drops solution (Active Comparator): 1 drop of NETILDEX™ (Netilmicin Sulfate 3mg/ml / Dexamethasone Disodium Phosphate 1mg/ml) eye drops solution immediately after the surgery then 1 drop four times a day (q.i.d.) from Day 1 until Day 14 after surgery.
  Bromfenac 0.9 mg/ml 1 drop twice daily (b.i.d.) for 3 days before cataract surgery.
  Interventions: Drug: NETILDEX™ eye drops solution

INTERVENTIONS:
Drug: NETILDEX™ ophthalmic gel — 1 drop of NETILDEX™ (Netilmicin Sulfate 3mg/ml / Dexamethasone Disodium Phosphate 1mg/ml) ophthalmic gel immediately after the surgery then 1 drop twice daily (b.i.d.) from Day 1 until Day 14 after surgery + 1 drop of XANTERGEL™ ophthalmic gel twice daily (b.i.d.) from Day 1 until Day 14 after surgery.
  Bromfenac 0.9 mg/ml 1 drop twice daily (b.i.d.) for 3 days before cataract surgery.
  Arms: NETILDEX™ ophthalmic gel
Drug: NETILDEX™ eye drops solution — 1 drop of NETILDEX™ (Netilmicin Sulfate 3mg/ml / Dexamethasone Disodium Phosphate 1mg/ml) eye drops solution immediately after the surgery then 1 drop four times a day (q.i.d.) from Day 1 until Day 14 after surgery.
  Bromfenac 0.9 mg/ml 1 drop twice daily (b.i.d.) for 3 days before cataract surgery.
  Arms: NETILDEX™ eye drops solution

SUMMARY:
Cataract is an ophthalmic disease that usually affects the elderly population. Cataract surgery with phaco-emulsification is now the most frequently performed intraocular surgical procedure in the developed world. However, differences in surgical technique impact the severity of surgical trauma and post-operative recovery. The amount of post-operative ocular pain and inflammation plays a significant role in the Patient's perception of the surgical success.

Several ophthalmic products have been studied in the management of post-surgery ocular inflammation and pain following cataract surgery. Corticosteroids are considered the gold standard for the treatment of ocular inflammation, and their most commonly used route of administration is the topical instillation as eye drops formulation.

After topical administration of Dexamethasone, the concentration in the anterior chamber increases and declines within hours, necessitating frequent daily instillations of eye drops for several weeks. This might be associated with compliance issues, particularly in elderly Patients or in individuals with disabilities. A pharmaceutical formulation allowing for a less frequent administration could therefore be an attractive alternative.

NETILDEX™ eye drops solution, containing Netilmicin Sulfate 4.55 mg (3mg/ml) and Dexamethasone Disodium Phosphate 1.32 mg (1mg/ml), is already available for Patients. A new ophthalmic gel, preservative-free formulation has been developed. This new formulation has been tested in pre-clinical animal studies and in a clinical trial. The new formulation contains Xanthan gum, a high molecular mass polysaccharide approved by the FDA in 1969 for food products. It is used in the product as viscosity enhancer and to give to the product pseudo-plastic characteristics and prolonged ocular retention time.

The purpose of this trial is to show that the administration of a reduced dose of NETILDEX ™ gel 2 times a day starting on the day of cataract extraction by means of phaco-emulsification and administered until 14 days after surgery is sufficient to obtain a non-inferior efficacy of the NETILDEX ™ eye drops solution administered 4 times a day for the same period.

DETAILED DESCRIPTION:
Cataract is an ophthalmic disease that usually affects the elderly population. Therapy is surgical and during the past decades, improvements in surgical techniques and instruments have dramatically increased the number of cataract extractions performed.

With improvements in surgical techniques, Patients' expectations have risen proportionally; however, differences in surgical technique impact the severity of surgical trauma and post-operative recovery. Cataract surgery with phaco-emulsification is now the most frequently performed intraocular surgical procedure in the developed world.

The amount of post-operative ocular pain and inflammation plays a significant role in the Patient's perception of the surgical success.

Ocular inflammation, commonly observed after cataract surgery, is associated with a breakdown of the blood-aqueous barrier (BAB) as a result of surgical trauma-induced prostaglandin production.

Anterior chamber ocular inflammation, clinically assessed as anterior chamber cell counts and flare, is also common following cataract surgery. However, post-surgery inflammation is frequently viewed as an acceptable risk that is largely outweighed by the numerous benefits of cataract surgery.

Advanced surgical techniques including phaco-emulsification, capsulorhexis, small clear corneal incisions, improved visco-elastics and foldable implants have helped to optimize post-surgery results and reduce surgical trauma. However, post-surgery inflammation may still occur and can lead to complications such as corneal edema, intra-ocular pressure (IOP) spikes, posterior capsule opacification and cystoid macular edema (CME).

The management of post-surgery inflammation is essential, both to ensure rapid recovery following surgery, and to prevent or decrease the potential for long-term complications, such as cystoid macular edema.

Several ophthalmic products have been studied for the management of post-surgery ocular inflammation and pain following cataract surgery. The two main treatments for ocular inflammation are topical corticosteroids or non-steroidal anti-inflammatory (NSAID) drugs.

Bromfenac is a potent inhibitor of the COX-2 enzyme and a highly lipophilic molecule that rapidly penetrates to produce early and sustained drug levels in all ocular tissues. Studies have shown that Bromfenac ophthalmic solution has equivalent efficacy to the other topical NSAIDs in reducing post-operative inflammation and controlling pain.

In order to decrease both intra-surgical and post-operative inflammation, it is now becoming commonplace to extend ophthalmic NSAID dosing to pre-operative use as well to reduce inflammation and minimize the risk of post-surgery complications in particular to prevent post-surgery cystoid macular edema.

Corticosteroids are considered the gold standard for the treatment of ocular inflammation, they are routinely used to control post-surgery ocular inflammation. The most commonly used route of administration of corticosteroid agents is the topical instillation as eye drops formulation. Steroids can be used as an additional prophylactic treatment in high-risk cases.

After topical administration of Dexamethasone, the concentration in the anterior chamber increases and declines within hours, necessitating frequent daily instillations of eye drops for several weeks. This might be associated with compliance issues, particularly in elderly Patients or in individuals with disabilities. A pharmaceutical formulation allowing for a less frequent administration could therefore be an attractive alternative.

Increase in intra-ocular pressure (IOP) is a concern after the use of corticosteroids, irrespective of the route of administration. Repeated use of topical steroids has been shown to induce reversible elevations in IOP, especially in eyes with glaucoma.

Although most of the Patients develop an increase in IOP after 3-6 weeks of treatment with topical steroids, some elevation of IOP can be found as early as the first or second week after initiation of topical instillation of steroids.

NETILDEX™ eye drops solution, containing Netilmicin Sulfate 4.55 mg (3mg/ml) and Dexamethasone Disodium Phosphate 1.32 mg (1mg/ml), is already available for Patients. A new ophthalmic gel, preservative-free formulation has been developed. This new formulation has been tested in pre-clinical animal studies and in a clinical trial. The new formulation contains Xanthan gum, a high molecular mass polysaccharide approved by the FDA in 1969 for food products and it is used in the product as viscosity enhancer and to give to the product pseudo-plastic characteristics and prolonged ocular retention time. Its usability in ophthalmic preparations is well known and another products containing Xanthan gum is currently available in the market (Timolol GFS, Falcon Pharmaceuticals, USA).

The penetration in the target tissue of Netilmicin and Dexamethasone contained in NETILDEX ™ eye drops and NETILDEX™ ophthalmic gel has been studied in a pre-clinical study in rabbits, which results suggest that the ophthalmic gel formulation increases the tissue bioavailability of both active principles.

A clinical study has been conducted in 63 healthy volunteers (21 per group) to establish the safety and ocular tolerability of NETILDEX ™ ophthalmic gel, in comparison with placebo and eye drop solution, administered q.i.d. (1 drop) over a period of 14 days . Both formulations were tolerated as placebo. A statistically significant difference between placebo and Dexamethasone/Netilmicin was observed, as expected, for intra-ocular pressure (IOP) values, however in none of the cases the IOP rising was clinically relevant.

The purpose of this trial is to show that the administration of a reduced dose of NETILDEX ™ gel 2 times a day starting on the day of cataract extraction by means of phaco-emulsification and administered until 14 days after surgery is sufficient to obtain a non-inferior efficacy of the NETILDEX ™ eye drops solution administered 4 times a day for the same period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Patients
2. Patients aged ≥ 40 years old
3. Patients undergoing cataract extraction surgery through phaco-emulsification and intra-ocular lens implantation
4. Patients with grade 2 or 3 according to LOCS III system for grading age-related cataract
5. Patients with transparent cornea (endothelial count in the limits for age but not lower than 1200 cells/mm2)
6. Patients understanding the nature of the study and providing their informed consent to participation
7. Patients willing and able to attend the visits and procedures foreseen by study protocol
8. Patients with negative Amsler Test at enrolment visit (V1)

Exclusion Criteria:

* Patients with medical history of ocular inflammation diseases, Herpes infections, iritis, uveitis or Sjogren's syndrome
* Patients who have been treated for external ocular infections within a month before the study enrolment (V1)
* Patients with cellularity in the anterior ocular chamber ≥ grade 2 (16-25 cells / field 1x1 mm)
* Patients with flare in the anterior ocular chamber ≥ grade 2 (moderate)
* Patients with at least one of the following concomitant ocular diseases: ocular infections, uveitis, iritis, iridociclitis, glaucoma, diabetic retinopathy, diabetes, maculopathy, shallow anterior chamber (based on Investigator's judgment)
* Patients with PEX Syndrome (Pseudo-exfoliation syndrome)
* Patients with poor mydriasis, basing on Investigator's judgment
* Patients with intra-ocular pressure > 24 mmHg
* Patients who have undergone surgery in the eye involved in the cataract extraction within the 12 months before the study enrolment (V1)
* Patients who have received corneal laser treatment in the eye involved in the cataract extraction within the 6 months before the study enrolment (V1)
* Patients with known or suspected allergy or hypersensitivity to ophthalmic preservatives, phenylacetic acid derivatives, aminoglycosides, Bromfenac, other NSAIDs, steroids
* Patients with traumatic cataract condition
* Patients who have been treated or are under treatment with alpha-blocking agents for more than 3 months before the study enrolment (V1)
* Patients who have received treatment with anti-histamines, decongestants, anti-inflammatory steroidal or non-steroidal (NSAID) drugs within the 15 days before the study enrolment (V1). Bromfenac, only, will be allowed for 3 days before cataract surgery
* Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment (V1)
* Patients receiving any ocular treatment, with the exception of artificial tears
* Female Patients who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical study and for three months later
* Female Patients of childbearing age (less than 24 months after the last menstrual cycle) who do not use adequate contraception *
* Monocle Patients
* Patients with epiretinal membrane as per OCT test at enrolment visit (V1)

  * Methods at low risk of contraceptive failure (less than 1% per year) when used consistently, including: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intra-uterine devices, abstinence or vasectomized partner. Contraception should be maintained until treatment discontinuation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Measurement of inflammation conditions in the anterior ocular chamber after cataract extraction through Slit Lamp and Bio-microscopy. | Throughout study completion, approximately 9 weeks.
  The measurement aims to demonstrate the efficacy of a reduced frequency of administration of NETILDEX™ ophthalmic gel, administered twice daily (b.i.d.), in comparison with NETILDEX™ eye drops solution, administered four times a day (q.i.d.), in the prevention of post-surgery inflammation after cataract extraction by means of phaco-emulsification.

SECONDARY OUTCOMES:
Evaluation of antibiotic efficacy based on the presence of detected microbial infections (positive ocular swabs and anti-biogram results, if any). | Within 24 hours after cataract surgery.
  The anti-biogram should be performed according to standard procedure at investigational sites, but including at least the test with Netilmicin and Cefuroxime.
Assessment of a potential variation in the intra-ocular pressure related to the use of the gel formulation compared to the eye-drops formulation, through its measurement before and after treatment. | Throughout study completion, approximately 9 weeks.
Evaluation of clinical signs and symptoms of ocular inflammation (other than flare and cellularity) through standard scoring systems. | Throughout study completion, approximately 9 weeks.
  In particular, attention will be focused on the evaluation in treated Patients of: degree of conjunctival hyperemia; lid/corneal edema; ocular discomfort.
Evaluation of visual acuity through standard measurement systems. | Throughout study completion, approximately 9 weeks.
Evaluation of the global tolerability of NETILDEX™ ophthalmic gel in treated Patients (by the Investigator), through a standard questionnaire. | Within 2 weeks after cataract surgery.
Evaluation of the safety of NETILDEX™ ophthalmic gel through the collection and evaluation of adverse events. | Throughout study completion, approximately 9 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Caporossi, MD, Prof., Principal Investigator — Policlinico Universitario A. Gemelli
Locations (7):
- Germany (2):
  - Klinikum Ernst von Bergmann Ophthalmologie, Potsdam
  - Augenklinik und Poliklinik Ophthalmologie, Würzburg
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Policlinico Universitario A. Gemelli, Roma
- Romania (2):
  - Centrul Medical Unirea, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrer A, Gerstmeyer K, Hirnschall N, Pesudovs K, Lundstrom M, Findl O. Impact of bilateral cataract surgery on vision-related activity limitations. J Cataract Refract Surg. 2013 May;39(5):680-5. doi: 10.1016/j.jcrs.2012.11.028. Epub 2013 Mar 25. PMID 23535380
- [Background] Porela-Tiihonen S, Kaarniranta K, Kokki H. Postoperative pain after cataract surgery. J Cataract Refract Surg. 2013 May;39(5):789-98. doi: 10.1016/j.jcrs.2013.03.012. PMID 23608571
- [Background] Monnet D, Tepenier L, Brezin AP. Objective assessment of inflammation after cataract surgery: comparison of 3 similar intraocular lens models. J Cataract Refract Surg. 2009 Apr;35(4):677-81. doi: 10.1016/j.jcrs.2008.12.021. PMID 19304088
- [Background] Goodman DF, Stark WJ, Gottsch JD. Complications of cataract extraction with intraocular lens implantation. Ophthalmic Surg. 1989 Feb;20(2):132-40. PMID 2648237
- [Background] Perry HD, Donnenfeld ED. An update on the use of ophthalmic ketorolac tromethamine 0.4%. Expert Opin Pharmacother. 2006 Jan;7(1):99-107. doi: 10.1517/14656566.7.1.99. PMID 16370927
- [Background] Sandoval HP, Fernandez de Castro LE, Vroman DT, Solomon KD. A review of the use of ketorolac tromethamine 0.4% in the treatment of post-surgical inflammation following cataract and refractive surgery. Clin Ophthalmol. 2007 Dec;1(4):367-71. PMID 19668513
- [Background] Alio JL, Sayans JA, Chipont E. Laser flare-cell measurement of inflammation after uneventful extracapsular cataract extraction and intraocular lens implantation. J Cataract Refract Surg. 1996;22 Suppl 1:775-9. doi: 10.1016/s0886-3350(96)80161-1. PMID 9279671
- [Background] Pande MV, Spalton DJ, Kerr-Muir MG, Marshall J. Postoperative inflammatory response to phacoemulsification and extracapsular cataract surgery: aqueous flare and cells. J Cataract Refract Surg. 1996;22 Suppl 1:770-4. doi: 10.1016/s0886-3350(96)80160-x. PMID 9279670
- [Background] Laurell CG, Zetterstrom C, Philipson B, Syren-Nordqvist S. Randomized study of the blood-aqueous barrier reaction after phacoemulsification and extracapsular cataract extraction. Acta Ophthalmol Scand. 1998 Oct;76(5):573-8. doi: 10.1034/j.1600-0420.1998.760512.x. PMID 9826042
- [Background] El-Harazi SM, Feldman RM. Control of intra-ocular inflammation associated with cataract surgery. Curr Opin Ophthalmol. 2001 Feb;12(1):4-8. doi: 10.1097/00055735-200102000-00002. PMID 11150074
- [Background] Rotsos TG, Moschos MM. Cystoid macular edema. Clin Ophthalmol. 2008 Dec;2(4):919-30. doi: 10.2147/opth.s4033. PMID 19668445
- [Background] Gulkilik G, Kocabora S, Taskapili M, Engin G. Cystoid macular edema after phacoemulsification: risk factors and effect on visual acuity. Can J Ophthalmol. 2006 Dec;41(6):699-703. doi: 10.3129/i06-062. PMID 17224950
- [Background] Cho H, Wolf KJ, Wolf EJ. Management of ocular inflammation and pain following cataract surgery: focus on bromfenac ophthalmic solution. Clin Ophthalmol. 2009;3:199-210. doi: 10.2147/opth.s4806. Epub 2009 Jun 2. PMID 19668566
- [Background] Rajpal RK, Ross B, Rajpal SD, Hoang K. Bromfenac ophthalmic solution for the treatment of postoperative ocular pain and inflammation: safety, efficacy, and patient adherence. Patient Prefer Adherence. 2014 Jun 25;8:925-31. doi: 10.2147/PPA.S46667. eCollection 2014. PMID 25028541
- [Background] Korenfeld MS, Silverstein SM, Cooke DL, Vogel R, Crockett RS; Difluprednate Ophthalmic Emulsion 0.05% (Durezol) Study Group. Difluprednate ophthalmic emulsion 0.05% for postoperative inflammation and pain. J Cataract Refract Surg. 2009 Jan;35(1):26-34. doi: 10.1016/j.jcrs.2008.09.024. PMID 19101421
- [Background] Lorenz K, Dick B, Jehkul A, Auffahrt GU. Inflammatory response after phacoemulsification treated with 0.5% prednisolone acetate or vehicle. Graefes Arch Clin Exp Ophthalmol. 2008 Nov;246(11):1617-22. doi: 10.1007/s00417-008-0908-2. Epub 2008 Aug 26. PMID 18726610
- [Background] Comstock TL, Paterno MR, Singh A, Erb T, Davis E. Safety and efficacy of loteprednol etabonate ophthalmic ointment 0.5% for the treatment of inflammation and pain following cataract surgery. Clin Ophthalmol. 2011;5:177-86. doi: 10.2147/OPTH.S16832. Epub 2011 Feb 10. PMID 21383946
- [Background] McGhee CN, Dean S, Danesh-Meyer H. Locally administered ocular corticosteroids: benefits and risks. Drug Saf. 2002;25(1):33-55. doi: 10.2165/00002018-200225010-00004. PMID 11820911
- [Background] Sanders DR, Kraff M. Steroidal and nonsteroidal anti-inflammatory agents. Effect on postsurgical inflammation and blood-aqueous humor barrier breakdown. Arch Ophthalmol. 1984 Oct;102(10):1453-6. doi: 10.1001/archopht.1984.01040031173012. PMID 6385931
- [Background] Corbett MC, Hingorani M, Boulton JE, Shilling JS. Subconjunctival betamethasone is of benefit after cataract surgery. Eye (Lond). 1993;7 ( Pt 6):744-8. doi: 10.1038/eye.1993.173. PMID 8119423
- [Background] Watson D, Noble MJ, Dutton GN, Midgley JM, Healey TM. Penetration of topically applied dexamethasone alcohol into human aqueous humor. Arch Ophthalmol. 1988 May;106(5):686-7. doi: 10.1001/archopht.1988.01060130748037. PMID 3358736
- [Background] Winfield AJ, Jessiman D, Williams A, Esakowitz L. A study of the causes of non-compliance by patients prescribed eyedrops. Br J Ophthalmol. 1990 Aug;74(8):477-80. doi: 10.1136/bjo.74.8.477. PMID 2390523
- [Background] ARMALY MF. EFFECT OF CORTICOSTEROIDS ON INTRAOCULAR PRESSURE AND FLUID DYNAMICS. I. THE EFFECT OF DEXAMETHASONE IN THE NORMAL EYE. Arch Ophthalmol. 1963 Oct;70:482-91. doi: 10.1001/archopht.1963.00960050484010. No abstract available. PMID 14078870
- [Background] BECKER B, MILLS DW. CORTICOSTEROIDS AND INTRAOCULAR PRESSURE. Arch Ophthalmol. 1963 Oct;70:500-7. doi: 10.1001/archopht.1963.00960050502012. No abstract available. PMID 14078872
- [Background] Bartlett JD, Woolley TW, Adams CM. Identification of high intraocular pressure responders to topical ophthalmic corticosteroids. J Ocul Pharmacol. 1993 Spring;9(1):35-45. doi: 10.1089/jop.1993.9.35. PMID 8463731
- [Background] Barry P, Cordovés L, Gardner S. ESCRS Guidelines for Prevention and Treatment of Endophthalmitis Following Cataract Surgery: Data, Dilemmas and Conclusions. The European Society for Cataract & Refractive Surgeons 2013